CLINICAL TRIAL: NCT04653714
Title: The Effects of Non-surgical Periodontal Therapy in Patients Indicated for Bariatric Surgery on the Periodontal and Systemic Inflammation Parameters: a Randomized Double Blinded Controlled Trial
Brief Title: The Effects of Non-surgical Periodontal Therapy in Patients Indicated for Bariatric Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ljubljana (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ULjubljana
Record Dates: First submitted 2020-10-23; First posted 2020-12-04 (Actual); Last update posted 2021-12-17 (Actual); Status verified 2021-12

CONDITIONS: Periodontitis; Obesity, Morbid; Bariatric Surgery Candidate
MeSH Terms: conditions — Periodontitis; Obesity, Morbid | interventions — Tooth Exfoliation; Root Planing

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Full mouth debridement (Experimental): Supragingival plaque/calculus removal and scaling and root planing
  Interventions: Procedure: Scaling and root planing
- Supragingival plaque/calculus removal (Sham Comparator): Supragingival plaque and calculus removal
  Interventions: Procedure: Scaling and root planing
- Probiotic lozenges (Experimental): Daily usage of probiotic lozenges
  Interventions: Device: Probiotic lozenges
- Placebo lozenges (Active Comparator): Daily usage of placebo lozenges
  Interventions: Device: Probiotic lozenges

INTERVENTIONS:
Procedure: Scaling and root planing — Patients with periodontitis in the test group will be treated by conventional non-surgical root debridement and in the control group by low-intensive supragingival plaque removal with mechanical brush and professional tooth paste only.
  Arms: Full mouth debridement; Supragingival plaque/calculus removal
Device: Probiotic lozenges — Patients with gingivitis in the test group will be treated with supragingival debridement and with probiotic lozenges with strains of Lactobacillus brevis and Lactobacillus plantarum once a day for 3 months and in the control group by low-intensive supragingival plaque removal, as a placebo treatment, and placebo probiotics lozenges.
  Arms: Placebo lozenges; Probiotic lozenges

SUMMARY:
By World Health Organization (WHO) definition overweight (body mass index (BMI) >24.9) and obesity (BMI >29.9) are defined as abnormal or excessive fat accumulation with many possible impacts on individual's health. Association between obesity and associated metabolic syndrome (obesity, hypertension, diabetes mellitus type 2 and dyslipidemia) and oral health has become clear from several studies that proved increased odds of obese patients for developing of caries-related pathologies and periodontal disease. Periodontal disease, a major cause of tooth loss in adults, is an inflammatory disease of periodontal tissue that is initiated by dental plaque bacteria and is modulated by the inflammatory-immune host response factors. Relation between periodontal disease and obesity is bi-directional, through sharing of several proposed local and systemic pathogenesis mechanisms. For treatment of obesity, bariatric surgery (BS) procedures are methods of choice, when other less invasive options fail. They are safe, cost-effective, improve overall health and increase life expectancy. There are several types of BS interventions and most commonly performed BS is laparoscopic sleeve gastrectomy and with second most often, Roux-en-Y gastric bypass. Studies on influence of BS on periodontal health showed diverse results, with some showing no effect, while others demonstrated an increase in the prevalence of periodontitis as well as a further deterioration of periodontal tissues after BS procedure. However, studies on the prevalence of gingivitis, a reversible plaque-induced inflammation of gingiva, and its progression to periodontitis in BS patients is lacking. Furthermore, dental and periodontal status are not routinely evaluated in patients before or after BS. To the best of our knowledge studies on the effect of periodontal therapy before BS are lacking.

DETAILED DESCRIPTION:
Obesity is becoming one of the mayor worldwide health problems due to increasing prevalence. In the Slovenia 63.4% of population are overweight (24.99 kg/m² < BMI < 29.99 kg/m²) and 28.6% are obese (BMI > 30 kg/m²). Obese patients have a predisposing factor of many chronic diseases including periodontal disease (PD). PD is an inflammatory disease of tooth supporting tissues that is initiated by dental plaque bacteria and modulated by the inflammatory-immune host response factors. Some of the causes for periodontitis in obese individuals are hyperinflammatory response, different fat metabolism and higher degree of insulin resistance. On the other hand, periodontitis is thought to have a negative effect on some obesity related comorbidities by rising systemic inflammation, increasing insulin resistance, lipid profile and endothelial function.

Several methods have been proposed for weight loss like dieting, physical exercise, pharmacologic treatment and surgical intervention. Bariatric surgery (BS) has been shown to be an effective weight loss strategy and is proposed as a frontline therapy for adult patients with severe obesity. The outcomes of bariatric surgery show decreased levels of pro-inflammatory markers such as Tumour Necrosis Factor alpha (TNF-α), interleukine-6 (IL6) and C-reactive protein (CRP) and therefore improvement of general inflammation status. Research papers observing association between BS and PD mostly advocate worsening of periodontal status and oral health as a complication of BS. Observational studies have shown that obese patients undergoing BS procedures have a high prevalence of periodontal disease and even though metabolic parameters are advancing to normal values after BS, inflammatory response to plaque bacteria in the gingiva is increased, with possible additional destruction of periodontal tissues. The reasons for high prevalence as well as deterioration after BS procedure is not completely understood. To the best of our knowledge, there are no interventional studies with non-surgical periodontal therapy that aim to lower PD progression after BS.

The aim is to investigate the influence of non-surgical periodontal therapy 1 month before BS in patients diagnosed with periodontitis and gingivitis on the level of reduction in local/systemic inflammatory and periodontal parameters. The second aim is to test whether implemented periodontal therapy has some impact on metabolic parameters and comorbidities of obesity after BS.

Participants will be selected in a randomized, interventional, blinded (examiner), prospective study, from 70 obese patients indicated for BS with criteria obesity class III (ITM over 40 kg/m2) and class I and II with obesity if related disease are present: diabetes mellitus type II, Hypertension, hyperlipidaemia, obstructive sleep apnea, articular pain, polycystic ovary syndrome. Patients will be recruited from Department of Abdominal Surgery, University Medical Centre Ljubljana, were BS procedure will be performed, and pre- and post-operative systemic and obesity related data will be collected. All relevant medical data will be taken from the records.

All the oral health intervention will be held at the Department for Oral Diseases and Periodontology, Dental Clinic, University Medical Centre Ljubljana. At the first visit general health, socioeconomic, dental information will be recorded by a questionnaire before surgical procedure. At the same time patients will undergo periodontal examination (number of the teeth, prosthetic rehabilitation status, full mouth plaque score (FMPS), full mouth bleeding score (FMBS), periodontal pocket depth (PPD), clinical attachment level (CAL), bleeding on probing (BOP), recession, furcation involvement, teeth mobility.

After oral examination, two study groups will be established (gingivitis n=30; and periodontitis patients n=40).

One month before scheduled BS periodontal therapy will be performed in all patients regarding their periodontal diagnosis (e.g. periodontitis or gingivitis) and previously predetermined randomisation to (test and control group) All included patients will be properly instructed and motivated for oral hygiene and fill out OHIP-14 questionnaire.

Patients with gingivitis in the test group (n=15) will be treated with supragingival debridement and with probiotic lozenges with strains of Lactobacillus brevis and Lactobacillus plantarum once a day for 3 months and in the control group (n=15) by low-intensive supragingival plaque removal, as a placebo treatment, and placebo probiotics lozenges.

Patients with periodontitis in the test group (n=20) will be treated by conventional non-surgical root debridement and in the control group (n=20), as a placebo treatment, by low-intensive supragingival plaque removal with mechanical brush and professional tooth paste only.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years patients undergoing BS (morbidly obese patients (obesity class III) and obese patients (class II and I) with obesity related comorbidities: diabetes mellites type II, Hypertension, hyperlipidaemia, obstructive sleep apnea, articular pain, polycystic ovary syndrome) from Department of Abdominal Surgery, University Medical Centre Ljubljana.
* ≥ 16 teeth present
* Diagnoses with periodontitis or gingivitis
* Singed consent

Exclusion Criteria:

* Antibiotic and periodontal therapy in previous 6 months
* The need of prophylactic antibiotic therapy
* Pregnant women, lactation
* Cancer and other serious chronic diseases (excluding metabolic syndrome) with known influence on periodontal health

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
Percentage of Bleeding on Probing (BOP) Sites | at 7 months after treatment
  Percentage of probing sites that bleed will be calcuated from fill mouth record

SECONDARY OUTCOMES:
Probing Pocket Depth (PPD) change | at 7 months post treatment
  Difference between the baseline and 7 months post-treatment PPD
Clinical Attachment Level (CAL) change | at 7 months post treatment
  Difference between the baseline and 7 months post-treatment CAL
C-reactive protein (CRP) | at 7 months post treatment
  CRP levels in the blood increase when there is a condition causing inflammation somewhere in the body.

OTHER OUTCOMES:
Oral Health Impact Profile (OHIP) -14 questionnaire | at 7 months post treatment
  OHIP is a standard oral health realted quality of life assessment tool

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Centre, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Colak D, Cmok Kucic A, Pintar T, Gaspirc B, Gaspersic R. Periodontal and systemic health of morbidly obese patients eligible for bariatric surgery: a cross-sectional study. BMC Oral Health. 2022 May 13;22(1):174. doi: 10.1186/s12903-022-02207-0. PMID 35562737